CLINICAL TRIAL: NCT00637975
Title: Randomized Phase II Trial Evaluating Activity and Tolerability of Fixed Dose of Oxycodone and Increasing Dose of Pregabalin Versus Increasing Dose of Oxycodone and Fixed Dose of Pregabalin for the Treatment of Oncological Neuropathic Pain
Brief Title: Oxycodone and Pregabalin for the Treatment of Oncological Neuropathic Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Associazione Progetto Oncologia UMAN.A (Other)
Collaborators: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Gabriella Farina, Fatebenefratelli and Ophtalmic Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEUROPAIN01; EudraCT Number 2007-005222-69
Record Dates: First submitted 2008-03-12; First posted 2008-03-18 (Estimated); Last update posted 2011-02-02 (Estimated); Status verified 2011-01

CONDITIONS: Cancer; Pain
Keywords: neuropathic pain; oxycodone; pregabalin; Patients with cancer and presenting a neuropathic pain
MeSH Terms: conditions — Neoplasms; Pain; Neuralgia | interventions — Oxycodone; Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): oxycodone 20 mg/day plus pregabalin at increasing dose starting from 50 mg/day for 15 days or until unacceptable toxicity develops
  Interventions: Drug: oxycodone; Drug: pregabalin
- B (Active Comparator): pregabalin 50 mg/day plus oxycodone at increasing dose starting from 20 mg/day. For 15 days or until unacceptable toxicity develops
  Interventions: Drug: oxycodone; Drug: pregabalin

INTERVENTIONS:
Drug: oxycodone — Arm A - 20 mg/day
  Arm B - increasing dose startnig at 20 mg/day
  For 15 days or until unacceptable toxicity develops.
Drug: pregabalin — Arm A - pregabalin at increasing dose starting from 50 mg/day
  Arm B - pregabalin 50 mg/day
  For 15 days or until unacceptable toxicity develops.

SUMMARY:
The aim of the study is to assess tolerability and activity of oxycodone and pregabalin in combination for the treatment of oncological neuropathic pain with two different strategies.

DETAILED DESCRIPTION:
Neuropathic pain is frequently diagnosed as a complication of cancer pain. While opioids are the mainstay of cancer pain management,their efficacy in neuropathic pain seems to be less then optimal,and adjuvant drugs, mainly anticonvulsants and antidepressants,are often combined with opioids in the analgesic regimen of patients with neuropathic cancer pain. This approach is suggested by well-established guidelines, but the analgesic benefit and the safety of pregabalin and oxycodone in combination is not yet documented.

The aim of this study is to assess the activity and tolerability of the addition of pregabalin to oxycodone in the treatment of patients with neuropathic pain due to neoplasm.

ELIGIBILITY:
Inclusion Criteria:

* instrumental and clinical diagnosis of every malignant neoplasm
* presence of pain with a neuropathic component in the opinion of the physician
* presence of pain >=4(NRS)
* PS ECOG <3
* written informed consent

Exclusion Criteria:

* serum creatinine >2mg/ml or creatinine clearance <40 ml/min
* mild or severe hepatic insufficiency
* iatrogenic neuropathy caused by chemotherapeutic agents
* previous allergic reactions to oxycodone and pregabalin
* pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2007-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Achievement of analgesia (decrease of at least 1/3 of pain intensity) assessed by NRS scale | within 15 days

SECONDARY OUTCOMES:
Pain control rate | within 15 days
Reduction of Break Through Pain number | within 15 days
Record of adverse events | within 15 days
Reduction of allodynia in patients presenting it at T0 | within 15 days
Patient satisfaction | within 15 days
Assessing whether COMT and mu blood polymorphisms are associated to response | within 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Gabriella Farina, MD, Principal Investigator — Fatebenefratelli and Ophtalmic Hospital
Locations (8):
- Italy (8):
  - Ospedale Fatebenefratelli, Benevento, Benevento
  - Ospedali Riuniti, Bergamo, Bergamo
  - Ospedale S. Orsola, Brescia, Brescia
  - Ospedale Serbelloni, Gorgonzola, Milano
  - Fatebenefratelli and Ophtalmic Hospital, Milan, Milano
  - Ospedale Civile di Legnano, Parabiago, Milano
  - Ospedale Fatebenefratelli, Roma, Roma
  - Ospedale Sacro Cuore, Negrar, Verona

REFERENCES:
- [Background] Merskey H, Bugduk N. Classification of chronic pain. Description of chronic pain. Description of chronic pain syndromes and definitions of chronic pain terms. Seattle: IASP, press 1994
- [Background] Negri E, Bettaglio R, Demartini L, Allegri M, Barbieri M, Miotti D, Paulin L, Buonocore M, Bonezzi C. [Validation of the Italian version of the "Neuropathic Pain Scale" and its clinical applications]. Minerva Anestesiol. 2002 Mar;68(3):95-104. Italian. PMID 11981518
- [Background] Riley J, Ross JR, Rutter D, Wells AU, Goller K, du Bois R, Welsh K. No pain relief from morphine? Individual variation in sensitivity to morphine and the need to switch to an alternative opioid in cancer patients. Support Care Cancer. 2006 Jan;14(1):56-64. doi: 10.1007/s00520-005-0843-2. Epub 2005 Jun 11. PMID 15952009
- [Background] Mucci-LoRusso P, Berman BS, Silberstein PT, Citron ML, Bressler L, Weinstein SM, Kaiko RF, Buckley BJ, Reder RF. Controlled-release oxycodone compared with controlled-release morphine in the treatment of cancer pain: a randomized, double-blind, parallel-group study. Eur J Pain. 1998;2(3):239-49. doi: 10.1016/s1090-3801(98)90020-9. PMID 15102384
- [Background] Bruera E, Belzile M, Pituskin E, Fainsinger R, Darke A, Harsanyi Z, Babul N, Ford I. Randomized, double-blind, cross-over trial comparing safety and efficacy of oral controlled-release oxycodone with controlled-release morphine in patients with cancer pain. J Clin Oncol. 1998 Oct;16(10):3222-9. doi: 10.1200/JCO.1998.16.10.3222. PMID 9779695
- [Background] Altier N, Dion D, Boulanger A, Choiniere M. Management of chronic neuropathic pain with methadone: a review of 13 cases. Clin J Pain. 2005 Jul-Aug;21(4):364-9. doi: 10.1097/01.ajp.0000125247.95213.53. PMID 15951657
- [Background] Gralow I. Cancer pain: an update of pharmacological approaches in pain therapy. Curr Opin Anaesthesiol. 2002 Oct;15(5):555-61. doi: 10.1097/00001503-200210000-00014. PMID 17019254
- [Background] Farrar JT, Portenoy RK. Neuropathic cancer pain: the role of adjuvant analgesics. Oncology (Williston Park). 2001 Nov;15(11):1435-42, 1445; discussion 1445, 1450-3. PMID 11758872
- [Background] Dirks J, Petersen KL, Rowbotham MC, Dahl JB. Gabapentin suppresses cutaneous hyperalgesia following heat-capsaicin sensitization. Anesthesiology. 2002 Jul;97(1):102-7. doi: 10.1097/00000542-200207000-00015. PMID 12131110
- [Background] Caraceni A, Zecca E, Bonezzi C, Arcuri E, Yaya Tur R, Maltoni M, Visentin M, Gorni G, Martini C, Tirelli W, Barbieri M, De Conno F. Gabapentin for neuropathic cancer pain: a randomized controlled trial from the Gabapentin Cancer Pain Study Group. J Clin Oncol. 2004 Jul 15;22(14):2909-17. doi: 10.1200/JCO.2004.08.141. PMID 15254060
- [Background] Mercadante S, Arcuri E, Tirelli W, Villari P, Casuccio A. Amitriptyline in neuropathic cancer pain in patients on morphine therapy: a randomized placebo-controlled, double-blind crossover study. Tumori. 2002 May-Jun;88(3):239-42. doi: 10.1177/030089160208800310. PMID 12195763
- [Background] Grond S, Zech D, Diefenbach C, Radbruch L, Lehmann KA. Assessment of cancer pain: a prospective evaluation in 2266 cancer patients referred to a pain service. Pain. 1996 Jan;64(1):107-114. doi: 10.1016/0304-3959(95)00076-3. PMID 8867252
- [Background] Portenoy RK, Foley KM, Inturrisi CE. The nature of opioid responsiveness and its implications for neuropathic pain: new hypotheses derived from studies of opioid infusions. Pain. 1990 Dec;43(3):273-286. doi: 10.1016/0304-3959(90)90025-9. PMID 1705692
- [Background] Chua KS, Reddy SK, Lee MC, Patt RB. Pain and loss of function in head and neck cancer survivors. J Pain Symptom Manage. 1999 Sep;18(3):193-202. doi: 10.1016/s0885-3924(99)00070-6. PMID 10517041
- [Background] Zech DFJ, Grond S, Lynch J, Hertel D, Lehmann KA. Validation of World Health Organization Guidelines for cancer pain relief: a 10-year prospective study. Pain. 1995 Oct;63(1):65-76. doi: 10.1016/0304-3959(95)00017-M. PMID 8577492
- [Background] Caraceni A. Clinicopathologic correlates of common cancer pain syndromes. Hematol Oncol Clin North Am. 1996 Feb;10(1):57-78. doi: 10.1016/s0889-8588(05)70327-0. PMID 8821560
- [Background] Elliott KJ. Taxonomy and mechanisms of neuropathic pain. Semin Neurol. 1994 Sep;14(3):195-205. doi: 10.1055/s-2008-1041078. No abstract available. PMID 7701120
- [Background] Kalso E. Oxycodone. J Pain Symptom Manage. 2005 May;29(5 Suppl):S47-56. doi: 10.1016/j.jpainsymman.2005.01.010. PMID 15907646
- [Background] Attal N, Cruccu G, Haanpaa M, Hansson P, Jensen TS, Nurmikko T, Sampaio C, Sindrup S, Wiffen P; EFNS Task Force. EFNS guidelines on pharmacological treatment of neuropathic pain. Eur J Neurol. 2006 Nov;13(11):1153-69. doi: 10.1111/j.1468-1331.2006.01511.x. PMID 17038030
- [Background] Bennett MI, Simpson KH. Gabapentin in the treatment of neuropathic pain. Palliat Med. 2004 Jan;18(1):5-11. doi: 10.1191/0269216304pm845ra. PMID 14982201
- [Background] Ross JR, Goller K, Hardy J, Riley J, Broadley K, A'hern R, Williams J. Gabapentin is effective in the treatment of cancer-related neuropathic pain: a prospective, open-label study. J Palliat Med. 2005 Dec;8(6):1118-26. doi: 10.1089/jpm.2005.8.1118. PMID 16351524
- [Background] Frampton JE, Foster RH. Pregabalin: in the treatment of postherpetic neuralgia. Drugs. 2005;65(1):111-8; discussion 119-20. doi: 10.2165/00003495-200565010-00011. PMID 15610058
- [Background] Davis MP. What is new in neuropathic pain? Support Care Cancer. 2007 Apr;15(4):363-72. doi: 10.1007/s00520-006-0156-0. Epub 2006 Nov 28. PMID 17131133
- [Background] Sonnett TE, Setter SM, Campbell RK. Pregabalin for the treatment of painful neuropathy. Expert Rev Neurother. 2006 Nov;6(11):1629-35. doi: 10.1586/14737175.6.11.1629. PMID 17144773
- [Background] Reyes-Gibby CC, Shete S, Rakvag T, Bhat SV, Skorpen F, Bruera E, Kaasa S, Klepstad P. Exploring joint effects of genes and the clinical efficacy of morphine for cancer pain: OPRM1 and COMT gene. Pain. 2007 Jul;130(1-2):25-30. doi: 10.1016/j.pain.2006.10.023. Epub 2006 Dec 6. PMID 17156920
- [Background] Simon R, Wittes RE, Ellenberg SS. Randomized phase II clinical trials. Cancer Treat Rep. 1985 Dec;69(12):1375-81. PMID 4075313
- [Background] Bruera E, Kuehn N, Miller MJ, Selmser P, Macmillan K. The Edmonton Symptom Assessment System (ESAS): a simple method for the assessment of palliative care patients. J Palliat Care. 1991 Summer;7(2):6-9. PMID 1714502
- [Background] Caraceni A, Mendoza TR, Mencaglia E, Baratella C, Edwards K, Forjaz MJ, Martini C, Serlin RC, de Conno F, Cleeland CS. A validation study of an Italian version of the Brief Pain Inventory (Breve Questionario per la Valutazione del Dolore). Pain. 1996 Apr;65(1):87-92. doi: 10.1016/0304-3959(95)00156-5. PMID 8826494
- [Derived] Garassino MC, Piva S, La Verde N, Spagnoletti I, Iorno V, Carbone C, Febbraro A, Bianchi A, Bramati A, Moretti A, Ganzinelli M, Marabese M, Gentili M, Torri V, Farina G. Randomised phase II trial (NCT00637975) evaluating activity and toxicity of two different escalating strategies for pregabalin and oxycodone combination therapy for neuropathic pain in cancer patients. PLoS One. 2013;8(4):e59981. doi: 10.1371/journal.pone.0059981. Epub 2013 Apr 5. PMID 23577077